CLINICAL TRIAL: NCT06876285
Title: Examination of the Effects of Wheelchair Treadmill Exercise and Conventional Wheelchair Exercises on Trunk Balance in Patients with Spinal Cord Injury
Brief Title: Effects of Wheelchair Treadmill and Conventional Exercises on Trunk Balance in Spinal Cord Injury Patients
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Sinem Yıldırım, M.Sc. physiotherapist, Ankara City Hospital Bilkent
Other Study IDs: TABED 1-24- 347
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
Keywords: postural balance; quality of life; functional indenpence
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group: Both groups will receive conventional physiotherapy, routinely administered in the clinic for 40 minutes, five days per week. Additional training sessions are planned for patients included in the study.
  Patients in the control group will receive at least 20 minutes of wheelchair propulsion training on a flat surface at least three days per week, in addition to the standard treatment. They will complete a total of 10 sessions within a maximum duration of four weeks.
- experimental group: Both groups will receive conventional physiotherapy, routinely administered in the clinic for 40 minutes, five days per week. Additional training sessions are planned for patients included in the study.
  Patients in the experimental group will participate in wheelchair treadmill training for at least 20 minutes per session, at least three days per week. They will complete a total of 10 treadmill training sessions within a maximum duration of four weeks.

SUMMARY:
This study aims to determine whether wheelchair treadmill exercises improve trunk balance and stability compared to conventional wheelchair exercises. Trunk balance is essential for mobility, transfers, and daily activities in individuals with spinal cord injury (SCI). The study includes individuals with SCI who use manual wheelchairs. Participants will be randomly assigned to: A control group performing conventional wheelchair exercises, an experimental group performing wheelchair treadmill exercises. Researchers will measure trunk balance, daily independence, wheelchair satisfaction, quality of life, and fear of falling. This research will help identify better rehabilitation methods for people with SCI.

This study is a prospective observational study. Regardless of whether the exercises are performed conventionally or using an alternative platform such as a wheelchair treadmill, all interventions included in the study are routine clinical practices. Patients whose treatment programs already adhere to the aforementioned procedures will be included in the study. In the Upper Extremity and Hand Rehabilitation Laboratory, where the wheelchair treadmill is available, patients with spinal cord injuries undergo a standardized rehabilitation program as part of routine clinical practice. This laboratory operates on a scheduled appointment basis.

After random allocation into groups, patients in the experimental group will be assessed at the beginning and end of the wheelchair treadmill therapy. Meanwhile, patients in the control group will be enrolled in the study before initiating wheelchair treadmill therapy. Once the data from the control group have been collected, these patients will also have the opportunity to receive wheelchair treadmill therapy.

DETAILED DESCRIPTION:
Our study is a prospective observational study. Regardless of whether the exercises are performed conventionally or using an alternative platform such as a wheelchair treadmill, all interventions included in the study are routine clinical practices. Patients whose treatment programs already adhere to the aforementioned procedures will be included in the study. In the Upper Extremity and Hand Rehabilitation Laboratory, where the wheelchair treadmill is available, patients with spinal cord injuries undergo a standardized rehabilitation program as part of routine clinical practice. This laboratory operates on a scheduled appointment basis.

After random allocation into groups, patients in the experimental group will be assessed at the beginning and end of the wheelchair treadmill therapy. Meanwhile, patients in the control group will be enrolled in the study before initiating wheelchair treadmill therapy. Once the data from the control group have been collected, these patients will also have the opportunity to receive wheelchair treadmill therapy.

The wheelchair treadmill to be utilized in the study is the h/p/cosmos saturn® 300/100 r model. The device includes two separate safety belts for the participant and the wheelchair, along with a wheelchair stabilizer equipped with three different locking mechanisms. Additionally, three emergency stop buttons located in different areas ensure maximum patient safety.

Treadmill exercises will be conducted at a submaximal level with a 0.7% incline. Heart rate will be monitored using a portable device. Regardless of whether the exercises are performed conventionally or on a treadmill, all exercises are part of routine clinical practice. Patients already receiving treatment in accordance with the aforementioned procedure will be included in the study. Participants will be randomly assigned to groups.

Data Quality and Management Procedures Patients admitted for inpatient treatment at the Spinal Cord Injury Rehabilitation Clinic of Ankara Bilkent City Hospital, who meet the inclusion criteria and voluntarily agree to participate in the study by reading and signing the informed consent form, will be included in the study. The medical status of all participants will be evaluated and recorded by the clinical research responsible physician. Exercise interventions will be carried out by two experienced physiotherapists working at the hospital. The patients' data will also be collected by these two physiotherapists.

Volunteers will be assessed at Ankara City Hospital Physical Therapy and Rehabilitation Hospital, within the Spinal Cord Injury Rehabilitation Neurophysiological Exercise Laboratory and the Upper Extremity and Hand Rehabilitation Laboratory, utilizing the treadmill available in the facility's sports hall.

A predefined data management plan will be implemented for missing, inconsistent, or erroneous data. Missing data will be identified and analyzed using statistical methods such as multiple imputation when necessary.

To ensure the integrity of data entry, regular audits and consistency checks will be performed by another physiotherapist involved in the study. To increase the reliability of the data, patient records and assessment reports will be cross-checked with the collected data. This will include comparisons made with electronic health records, paper-based case reports, and direct observation notes. All study procedures, including patient recruitment, data collection, data entry, data analysis, and reporting of adverse events, will be carried out according to predefined criteria.

Any adverse events or unexpected complications occurring during the study will be systematically documented and reported.

To determine the appropriate sample size, 10 patients per group will be included. Based on the obtained pilot data, a power analysis will be conducted using the G* Power program (version 3.0.10, Universität Düsseldorf, Düsseldorf, Germany).

For statistical analysis, descriptive statistics will be presented as the mean and standard deviation for numerical variables if the parametric assumptions are met, and as the median and minimum-maximum values if the parametric assumptions are not met. For categorical variables, frequency and percentage values will be reported. The statistical significance of differences between groups will be examined using the Independent Samples T-Test if parametric assumptions are met, and the Mann-Whitney U Test if parametric assumptions are not met. Analyses will be conducted with a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* SCI at the T6 level or below
* Classified as ASIA A or B
* Manual wheelchair user for at least four weeks
* Spinal stabilization achieved
* Voluntary consent to participate

Exclusion Criteria:

* Presence of osteoporosis
* Presence of cardiopulmonary disease
* Presence of a neurological condition other than SCI
* Presence of a musculoskeletal disorder affecting the joints or surrounding tissues
* Presence of orthostatic hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ankara bilkent city hospital
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Modified Functional Reach Test | 4 weeks
  During this test, the participant is seated on a chair with back support, with hips, knees, and feet positioned at 90-degree flexion and feet flat on the ground. A measuring tape is fixed to the wall at the level of the participant's acromion. The participant is instructed to bring their dominant arm to 90-degree flexion, and the initial measurement is recorded. The reference point for measurement is the styloid process of the ulna. Subsequently, the participant is asked to reach forward as far as possible. The contralateral hand is placed on the umbilicus to prevent compensatory stabilization.

SECONDARY OUTCOMES:
Trunk Control Test | 4 weeks
  This test evaluates both dynamic and static balance. It consists of 13 items, and participants are required to perform each activity three times, with the best score recorded. This validated and reliable scale assesses dynamic balance while performing upper extremity activities. Activities are scored between 0 and 2 (rolling movement is scored between 0 and 1). A high score indicates good trunk balance.
Spinal Cord Independence Measure | 4 weeks
  Spinal Cord Independence Measure has been developed to address three specific areas of function in patients with spinal cord injuries. It looks at self-care (feeding, grooming, bathing, and dressing), respiration and sphincter management, and a patient's mobility abilities (bed and transfers and indoors/outdoors).Scores range from 0-100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence. Each subscale score is evaluated within the 100-point scale (self-care: 0-20; respiration and sphincter management: 0-40; mobility: 0-40)
Quebec Assistive Technology User Satisfaction Assessment | 4 weeks
  Quebec Assistive Technology User Satisfaction Assessment is a 12-item questionnaire which assesses patients' satisfaction with assistive technology, including wheelchairs. Each item is rated on a six-point scale ranging from 'not at all satisfied' to 'very satisfied'. Eight items relate to the device and four items to service provision. Maximum score is 5, minimum score is 0. A high score indicates high satisfaction with the auxiliary equipment.
The 36-Item Short Form Survey | 4 weeks
  The 36-Item Short Form Survey will be utilized to assess quality of life. This questionnaire consists of 36 questions divided into eight subcategories: physical function, physical role limitations, pain, general health, vitality, social function, emotional role limitations, and mental health. Scores range from 0 (worst health) to 100 (best health).
Visual Analog Scale | 4 weeks
  Participants' fear of falling will be assessed using the Visual Analog Scale. The visual analog scale is a straight horizontal line with a fixed length of 100 mm. The extreme points are defined as the extreme limits of fear of falling and are directed from left (worst) to right (best). The patient marks the point on the line where he/she feels he/she perceives his/her current situation. The score of the visual analog scale is determined by measuring in millimeters from the left end of the line to the point marked by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No